CLINICAL TRIAL: NCT02487108
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase 3 Study to Evaluate the Analgesic Efficacy and Safety of Hydrocodone Bitartrate/Acetaminophen Immediate-Release Tablets (TV-46763) at Doses of 5.0 mg/325 mg, 7.5 mg/325 mg, and 10 mg/325 mg Every 4 to 6 Hours in Patients With Moderate to Severe Pain Following Bunionectomy
Brief Title: Study to Evaluate the Analgesic Efficacy and Safety of Hydrocodone Bitartrate/Acetaminophen Immediate-Release Tablets in Participants With Moderate to Severe Pain Following Bunionectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TV46763-CNS-30031
Record Dates: First submitted 2015-06-29; First posted 2015-07-01 (Estimated); Results first posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Hydrocodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Participants will receive placebo matching to TV46763 (hydrocodone bitartrate/acetaminophen) immediate release (IR) tablets for 48 hours (every 4 to 6 hours) on Days 1, 2, and 3 during the inpatient treatment period. Participants will continue to take the same treatment daily, every 4 to 6 hours after discharge on Day 3, over a 10-day (±1 day) outpatient treatment period.
  Interventions: Drug: Placebo
- TV-46763 5.0 mg/325 mg (Experimental): Participants will receive TV46763 (hydrocodone bitartrate/acetaminophen) 5.0 mg/325 mg IR tablets for 48 hours (every 4 to 6 hours) on Days 1, 2, and 3 during the inpatient treatment period. Participants will continue to take the same treatment daily, every 4 to 6 hours after discharge on Day 3, over a 10-day (±1 day) outpatient treatment period.
  Interventions: Drug: TV-46763
- TV-46763 7.5 mg/325 mg (Experimental): Participants will receive TV46763 (hydrocodone bitartrate/acetaminophen) 7.5 mg/325 mg IR tablets for 48 hours (every 4 to 6 hours) on Days 1, 2, and 3 during the inpatient treatment period. Participants will continue to take the same treatment daily, every 4 to 6 hours after discharge on Day 3, over a 10-day (±1 day) outpatient treatment period.
  Interventions: Drug: TV-46763
- TV-46763 10.0 mg/325 mg (Experimental): Participants will receive TV46763 (hydrocodone bitartrate/acetaminophen) 10.0 mg/325 mg IR tablets for 48 hours (every 4 to 6 hours) on Days 1, 2, and 3 during the inpatient treatment period. Participants will continue to take the same treatment daily, every 4 to 6 hours after discharge on Day 3, over a 10-day (±1 day) outpatient treatment period.
  Interventions: Drug: TV-46763

INTERVENTIONS:
Drug: TV-46763 — TV-46763 will be administered per dose and schedule specified in the arm description.
  Other Names: Hydrocodone bitartrate/acetaminophen IR tablets
  Arms: TV-46763 10.0 mg/325 mg; TV-46763 5.0 mg/325 mg; TV-46763 7.5 mg/325 mg
Drug: Placebo — Placebo matching to TV-46763 will be administered per schedule specified in the arm description.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the analgesic efficacy of hydrocodone bitartrate/acetaminophen immediate-release tablets at doses of 5.0 milligrams (mg)/325 mg, 7.5 mg/325 mg, and 10 mg/325 mg every 4 to 6 hours compared with placebo in treating participants with moderate to severe pain following bunionectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 to 75 years, inclusive.
2. Participants who are scheduled to undergo a primary unilateral first metatarsal Austin bunionectomy with distal osteotomy and internal fixation without any collateral procedures (ie, uncomplicated procedure).
3. Participants who according to the American Society of Anesthesiologists Physical Status (PS) classification system are classified PS-1 (normal, healthy participant) or PS-2 (mild systemic disease).
4. The participant is able to speak English and is willing to provide written informed consent, including a written opioid agreement, to participate in the study.
5. The participant has a body mass index (BMI) between 18.0 and 33.0 kg/m2 (inclusive) at the time of screening.
6. The participant is in generally good health as determined by a medical history, medical examination, ECG, serum chemistry, hematology, urinalysis, and serology.
7. Women of childbearing potential (not surgically sterile or 2 years postmenopausal) must use a medically acceptable method of contraception and must agree to continue use of this method for the duration of the study and for 30 days after discontinuation of the study drug, unless they have exclusively same-sex partners. Acceptable methods of contraception include intrauterine device (IUD) known to have a failure rate of less than 1% per year, hormonal contraceptive (oral, implanted, transdermal, or injected), and barrier method with spermicide, abstinence, and partner vasectomy.

   NOTE: A woman will be considered surgically sterile if she has had a tubal ligation, hysterectomy, bilateral salpingo-oophorectomy or bilateral oophorectomy, or hysterectomy with bilateral salpingo-oophorectomy.
8. The participant, if a man, is surgically sterile, or, if capable of producing offspring, is currently using a medically acceptable method of contraception and agrees to continue use of this method for the duration of the study (and for 90 days after taking the last dose of the study drug because of the possible effects on spermatogenesis), unless he has exclusively same-sex partners. Acceptable methods of contraception include abstinence, barrier method with spermicide, female partner's use of steroidal hormonal contraceptive (oral, implanted, transdermal, or injected) in conjunction with a barrier method, female partner's use of an IUD known to have a failure rate of less than 1% per year, or if his female partner is surgically sterile or 2 years postmenopausal. In addition, male participants may not donate sperm for the duration of the study and for 90 days after taking study drug.
9. The participant must be willing and able to comply with study restrictions and to remain at the clinic for the required duration during the study, and willing to return to the clinic for the follow-up evaluation as specified in this protocol.
10. The participant must not participate in any other study involving an investigational agent while enrolled in the present study.
11. The participant must report a pain intensity score of ≥4 on an 11-point NPRS-11 within 9 hours after stopping postsurgical analgesia and immediately before randomization.
12. The participant should be free of any surgical or anesthetic complications after the surgery, which is to be performed using the intraoperative anesthetic regimen and the postoperative analgesic regimen that was followed appropriately without deviations that would confound analgesic assessments after receipt of the investigational product.

Exclusion Criteria:

1. The participant has a chronic pain condition, excluding bunion pain that requires taking opioid analgesics within 30 days prior to surgery or use of non-opioid analgesics (acetylsalicylic acid, acetaminophen, nonsteroidal anti-inflammatory drugs) within 24 hours prior to surgery. Stable therapy of >30 days for acetylsalicylic acid (up to 81 mg/day) is allowed as cardiovascular prophylaxis.
2. Use of glucocorticoids (except nasal corticosteroid sprays and/or topical corticosteroids) for any condition within 6 months before study drug administration.
3. The participant uses any nonpharmacologic pain management techniques (eg, physical techniques, physiotherapy, massage therapy, acupuncture, biofeedback, and/or psychological support) and is unable or unwilling to discontinue prior to randomization (or study start).
4. The participant has any other medical or psychiatric condition or is receiving concomitant medication/therapy that would, in the opinion of the investigator, compromise the participant's safety, compliance with the study protocol procedures, or collection of data.
5. The participant has a clinically significant abnormality in the physical examination and/or clinical laboratory test values.
6. The participant is a pregnant or lactating woman. (Any woman becoming pregnant during the study will be withdrawn from the study.)
7. The participant has used an investigational drug within 1 month before the screening visit.
8. The participant is participating any currently ongoing research study.
9. The participant has any disorder that may interfere with gastrointestinal (GI) drug absorption (eg, gastric bypass surgery, lap band, malabsorption syndrome, and inflammatory bowel disease) or other condition that may have an effect on participant safety or efficacy aspects of participation in the opinion of the investigator.
10. The participant is allergic to or has had a serious reaction to hydrocodone or other opioids, acetaminophen, ropivacaine, lidocaine, ketorolac, ibuprofen, propofol, or any of the drugs required by the study protocol.
11. The participant has a recent history (within 5 years) or current evidence of alcohol or other substance abuse, with the exception of nicotine.
12. The participant has a positive urine drug screen (UDS) for cocaine, marijuana, opioids, amphetamines, methamphetamines, benzodiazepines, barbiturates, and/or methadone, unless explained by the use of prescription medication.
13. The participant has a history of suicidality as assessed by participant medical history and/or the C-SSRS.
14. The participant is expected to have elective surgery during the study other than a bunionectomy.
15. The participant has a history of malignancy within 5 years (except for treated basal cell carcinoma).
16. The participant has a positive test result for hepatitis B surface antigen or antibodies to hepatitis C, or known or tested positive for human immunodeficiency virus.
17. The participant has received a monoamine oxidase inhibitor (MAOI) within 14 days before the first dose of study drug.
18. The investigator believes that the participant is not suitable for the study for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 569 (Actual)
Dates: Start 2015-08-11 (Actual); Primary Completion 2016-03-30 (Actual); Study Completion 2016-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (8):
- United States (8):
  - Teva Investigational Site 13510, Phoenix, Arizona
  - Teva Investigational Site 13173, Anaheim, California
  - Teva Investigational Site 13174, Bakersfield, California
  - Teva Investigational Site 13170, Pasadena, California
  - Teva Investigational Site 13169, Pasadena, Maryland
  - Teva Investigational Site 13172, San Antonio, Texas
  - Teva Investigational Site 13171, Salt Lake City, Utah
  - Teva Investigational Site 13511, St. George, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo matched to TV46763 (hydrocodone bitartrate/acetaminophen) immediate release (IR) tablets for 48 hours (every 4 to 6 hours) on Days 1, 2, and 3 during the inpatient treatment period. Participants continued to take the same treatment daily, every 4 to 6 hours after discharge on Day 3, over a 10-day (±1 day) outpatient treatment period.
- TV-46763 5.0 mg/325 mg: Participants received TV46763 (hydrocodone bitartrate/acetaminophen) 5.0 milligrams (mg)/325 mg IR tablets for 48 hours (every 4 to 6 hours) on Days 1, 2, and 3 during the inpatient treatment period. Participants continued to take the same treatment daily, every 4 to 6 hours after discharge on Day 3, over a 10-day (±1 day) outpatient treatment period.
- TV-46763 7.5 mg/325 mg: Participants received TV46763 (hydrocodone bitartrate/acetaminophen) 7.5 mg/325 mg IR tablets for 48 hours (every 4 to 6 hours) on Days 1, 2, and 3 during the inpatient treatment period. Participants continued to take the same treatment daily, every 4 to 6 hours after discharge on Day 3, over a 10-day (±1 day) outpatient treatment period.
- TV-46763 10.0 mg/325 mg: Participants received TV46763 (hydrocodone bitartrate/acetaminophen) 10.0 mg/325 mg IR tablets for 48 hours (every 4 to 6 hours) on Days 1, 2, and 3 during the inpatient treatment period. Participants continued to take the same treatment daily, every 4 to 6 hours after discharge on Day 3, over a 10-day (±1 day) outpatient treatment period.
Period: Overall Study
Arm/Group | Placebo | TV-46763 5.0 mg/325 mg | TV-46763 7.5 mg/325 mg | TV-46763 10.0 mg/325 mg
Started | 142 | 142 | 143 | 142
Received at Least 1 Dose of Study Drug | 142 | 142 | 141 | 142
Completed | 126 | 126 | 117 | 131
Not Completed | 16 | 16 | 26 | 11
Not completed — Adverse Event | 1 | 6 | 12 | 6
Not completed — Withdrawal by Subject | 8 | 5 | 5 | 0
Not completed — Non-compliance to study medication | 3 | 2 | 5 | 4
Not completed — Protocol Violation | 1 | 1 | 2 | 0
Not completed — Non-compliance to study procedures | 0 | 0 | 0 | 1
Not completed — Other than specified | 3 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis set included all randomized participants.
Groups:
- Placebo: Participants received placebo matched to TV46763 (hydrocodone bitartrate/acetaminophen) IR tablets for 48 hours (every 4 to 6 hours) on Days 1, 2, and 3 during the inpatient treatment period. Participants continued to take the same treatment daily, every 4 to 6 hours after discharge on Day 3, over a 10-day (±1 day) outpatient treatment period.
- TV-46763 5.0 mg/325 mg: Participants received TV46763 (hydrocodone bitartrate/acetaminophen) 5.0 mg/325 mg IR tablets for 48 hours (every 4 to 6 hours) on Days 1, 2, and 3 during the inpatient treatment period. Participants continued to take the same treatment daily, every 4 to 6 hours after discharge on Day 3, over a 10-day (±1 day) outpatient treatment period.
- Total: Total of all reporting groups
Arm/Group | Placebo | TV-46763 5.0 mg/325 mg | TV-46763 7.5 mg/325 mg | TV-46763 10.0 mg/325 mg | Total
Number analyzed (Participants) | 142 | 142 | 143 | 142 | 569
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (14.39) | 45.8 (14.45) | 44.9 (13.87) | 46.2 (13.94) | 46.1 (14.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 124 | 125 | 113 | 481
  Male | 23 | 18 | 18 | 29 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 35 | 49 | 47 | 171
  Not Hispanic or Latino | 102 | 107 | 94 | 94 | 397
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 111 | 102 | 104 | 107 | 424
  Black | 24 | 30 | 29 | 26 | 109
  Asian | 4 | 8 | 7 | 5 | 24
  American Indian or Alaskan Native | 1 | 1 | 0 | 1 | 3
  Native Hawaiian or Pacific Islander | 0 | 1 | 0 | 1 | 2
  Other | 2 | 0 | 3 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Summed Pain Intensity Difference (SPID) Score Calculated Over the First 48 Hours (SPID48) After the First Dose of Study Drug on an 11-Point Numerical Pain Rating Scale (NPRS-11)
Description: The SPID48 was calculated as the time-weighted sum of pain intensity difference (PID) at each time point over 48 hours. The SPID48 was based on the NPRS-11, which is an 11-point Likert-type scale in which 0 means no pain and 10 means the most intense pain imaginable. Least square (LS) mean was calculated using an analysis of covariance (ANCOVA) with treatment and center as factors and the baseline pain intensity score as a covariate. Multiple imputation method was used to handle missing data.
Time Frame: 48 hours
Population: The full analysis set (FAS) included all randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TV-46763 5.0 mg/325 mg | TV-46763 7.5 mg/325 mg | TV-46763 10.0 mg/325 mg
Number analyzed (Participants) | 142 | 142 | 141 | 142
units on a scale | 76.5 (6.92) | 115.4 (6.92) | 120.5 (6.91) | 129.9 (6.88)
Statistical Analysis 1: Comparison: Placebo vs TV-46763 5.0 mg/325 mg; Analysis was performed using ANCOVA with treatment and center as factors and the baseline pain intensity score as a covariate; Test type: Other; p < 0.001, ANCOVA; LS Mean Difference = 38.9, 95% CI 2-sided [19.931 to 57.855]
Statistical Analysis 2: Comparison: Placebo vs TV-46763 7.5 mg/325 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.001, ANCOVA; LS Mean Difference = 44.0, 95% CI 2-sided [25.122 to 62.881]
Statistical Analysis 3: Comparison: Placebo vs TV-46763 10.0 mg/325 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.001, ANCOVA; LS Mean Difference = 53.4, 95% CI 2-sided [34.589 to 72.282]

2. Secondary Outcome: SPID Scores Over the Intervals During the First 36 Hours Following the First Dose of Study Drug
Description: The SPID was calculated as the time-weighted sum of PID at each time point over the intervals during the first 36 hours. The SPID was based on the NPRS-11, which is an 11-point Likert-type scale in which 0 means no pain and 10 means the most intense pain imaginable. LS mean was calculated using ANCOVA with treatment and center as factors and the baseline pain intensity score as a covariate. Multiple imputation method was used to handle missing data.
Time Frame: 0 to 6, 0 to 12, 0 to 24, and 0 to 36 hours
Population: The FAS included all randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TV-46763 5.0 mg/325 mg | TV-46763 7.5 mg/325 mg | TV-46763 10.0 mg/325 mg
Number analyzed (Participants) | 142 | 142 | 141 | 142
units on a scale
  SPID 0-6 | 3.7 (0.87) | 8.3 (0.87) | 8.3 (0.87) | 9.1 (0.88)
  SPID 0-12 | 6.4 (1.78) | 15.8 (1.77) | 16.5 (1.76) | 19.1 (1.78)
  SPID 0-24 | 21.1 (3.55) | 43.9 (3.53) | 44.5 (3.53) | 50.9 (3.53)
  SPID 0-36 | 44.2 (5.26) | 78.2 (5.26) | 81.1 (5.22) | 88.2 (5.22)

3. Secondary Outcome: Pain Intensity Difference (PID) Scores
Description: The PID was based on the NPRS-11, which is an 11-point Likert-type scale in which 0 means no pain and 10 means the most intense pain imaginable. PID was calculated at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, and 6 hours after the first dose of study drug. LS mean was calculated using ANCOVA with treatment and center as factors and the baseline pain intensity score as a covariate. Multiple imputation method was used to handle missing data.
Time Frame: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, and 6 hours
Population: The FAS included all randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TV-46763 5.0 mg/325 mg | TV-46763 7.5 mg/325 mg | TV-46763 10.0 mg/325 mg
Number analyzed (Participants) | 142 | 142 | 141 | 142
units on a scale
  0.25 hour | 0.1 (0.11) | 0.2 (0.11) | 0.1 (0.11) | 0.0 (0.11)
  0.5 hour | 0.5 (0.15) | 0.5 (0.15) | 0.8 (0.15) | 0.5 (0.15)
  0.75 hour | 0.6 (0.17) | 0.9 (0.17) | 1.4 (0.17) | 1.1 (0.17)
  1 hour | 0.7 (0.19) | 1.4 (0.19) | 1.8 (0.19) | 1.5 (0.19)
  1.5 hours | 0.8 (0.21) | 1.6 (0.21) | 2.2 (0.21) | 2.0 (0.21)
  2 hours | 0.8 (0.20) | 1.9 (0.20) | 2.2 (0.20) | 2.1 (0.20)
  3 hours | 1.0 (0.20) | 1.8 (0.20) | 1.7 (0.20) | 1.7 (0.20)
  4 hours | 0.7 (0.19) | 1.3 (0.19) | 1.0 (0.19) | 1.3 (0.19)
  5 hours | 0.6 (0.19) | 1.4 (0.19) | 1.2 (0.19) | 1.6 (0.19)
  6 hours | 0.4 (0.19) | 1.3 (0.19) | 1.3 (0.19) | 1.7 (0.19)

4. Secondary Outcome: Time to Peak PID
Description: Time to peak PID after the first dose of study drug but before the second dose of study drug was calculated. Kaplan-Meier method was used to calculate the data. Multiple imputation method was used to handle missing pain intensity scores at scheduled time points.
Time Frame: Within 6 hours
Population: The FAS included all randomized participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Placebo | TV-46763 5.0 mg/325 mg | TV-46763 7.5 mg/325 mg | TV-46763 10.0 mg/325 mg
Number analyzed (Participants) | 142 | 142 | 141 | 142
hours | 3.0 [2.02 to 3.03] | 2.0 [1.53 to 2.02] | 1.53 [1.52 to 2.01] | 2.0 [1.53 to 2.02]

5. Secondary Outcome: Number of Participants With a 30% Reduction in Pain Intensity Measured Using NPRS-11 Scores
Description: Number of participants with a 30% reduction in NPRS-11 scores was reported at 6, 12, 24, and 48 hours after the first dose of study drug.
Time Frame: 2, 4, 6, 12, 24, and 48 hours
Population: The FAS included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TV-46763 5.0 mg/325 mg | TV-46763 7.5 mg/325 mg | TV-46763 10.0 mg/325 mg
Number analyzed (Participants) | 142 | 142 | 141 | 142
Participants
  2 hours | 41 | 71 | 76 | 83
  4 hours | 39 | 44 | 41 | 60
  6 hours | 32 | 56 | 51 | 66
  12 hours | 38 | 55 | 54 | 76
  24 hours | 67 | 83 | 80 | 91
  48 hours | 86 | 96 | 92 | 100

6. Secondary Outcome: Number of Participants With a 50% Reduction in Pain Intensity Measured Using NPRS-11 Scores
Description: Number of participants with a 50% reduction in NPRS-11 scores was reported at 6, 12, 24, and 48 hours after the first dose of study drug.
Time Frame: 2, 4, 6, 12, 24, and 48 hours
Population: The FAS included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TV-46763 5.0 mg/325 mg | TV-46763 7.5 mg/325 mg | TV-46763 10.0 mg/325 mg
Number analyzed (Participants) | 142 | 142 | 141 | 142
Participants
  2 hours | 27 | 52 | 63 | 63
  4 hours | 20 | 29 | 28 | 40
  6 hours | 18 | 40 | 39 | 45
  12 hours | 22 | 33 | 31 | 52
  24 hours | 46 | 66 | 63 | 75
  48 hours | 73 | 75 | 79 | 90

7. Secondary Outcome: Time to Onset of Perceptible Pain Relief (PPR)
Description: Time to perceptible pain relief (PPR) (i.e., onset of pain relief) after the first dose of study drug was calculated using the stopwatch technique. The PPR stopwatch was started immediately after administration of the first dose of study drug (time zero [T0]) and it was given to the participant with the instructions to stop the stopwatch when he or she first perceived pain relief (time to perceptible relief). Kaplan-Meier method was used to calculate the data.
Time Frame: Day 1
Population: The FAS included all randomized participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: hour
Arm/Group | Placebo | TV-46763 5.0 mg/325 mg | TV-46763 7.5 mg/325 mg | TV-46763 10.0 mg/325 mg
Number analyzed (Participants) | 142 | 142 | 141 | 142
hour | 0.8 [0.50 to 1.23] | 0.5 [0.38 to 0.75] | 0.5 [0.47 to 0.68] | 0.6 [0.48 to 0.77]

8. Secondary Outcome: Time to Onset of Meaningful Pain Relief (MPR)
Description: Time to meaningful pain relief (MPR) after the first dose of study drug was calculated using the stopwatch technique. The MPR stopwatch was started immediately after administration of the first dose of study drug (time zero [T0]). The stopwatch was given to the participant with the instructions to stop the stopwatch when he or she first experienced meaningful pain relief (time to meaningful relief). Kaplan-Meier method was used to calculate the data.
Time Frame: Day 1
Population: The FAS included all randomized participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: hour
Arm/Group | Placebo | TV-46763 5.0 mg/325 mg | TV-46763 7.5 mg/325 mg | TV-46763 10.0 mg/325 mg
Number analyzed (Participants) | 142 | 142 | 141 | 142
hour | NA [NA to NA] — Due to smaller number of participants with an event, median and upper and lower limit of 95% confidence interval (CI) could not be calculated. | 1.9 [1.43 to 3.02] | 1.3 [1.00 to 2.22] | 1.8 [1.25 to NA] — Due to smaller number of participants with an event, upper limit of 95% CI could not be calculated.

9. Secondary Outcome: Total Rescue Medication Use (Number of Tablets Used)
Description: Total rescue medication (oral nonprescription ibuprofen) use (number of tablets used) over 6, 12, 24, and 48 hours after the first dose of study drug was calculated.
Time Frame: 6, 12, 24, and 48 hours
Population: The FAS included all randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: tablets
Arm/Group | Placebo | TV-46763 5.0 mg/325 mg | TV-46763 7.5 mg/325 mg | TV-46763 10.0 mg/325 mg
Number analyzed (Participants) | 142 | 142 | 141 | 142
tablets
  Total rescue medication use over 6 hours | 1.2 (0.07) | 0.8 (0.07) | 0.7 (0.07) | 0.6 (0.07)
  Total rescue medication use over 12 hours | 2.0 (0.10) | 1.4 (0.10) | 1.4 (0.10) | 1.1 (0.10)
  Total rescue medication use over 24 hours | 3.0 (0.13) | 2.1 (0.13) | 1.9 (0.13) | 1.6 (0.13)
  Total rescue medication use over 48 hours | 4.4 (0.22) | 2.9 (0.21) | 2.6 (0.21) | 2.1 (0.22)

10. Secondary Outcome: Number of Participants Taking Rescue Medication
Description: Number of participants taking rescue medication (oral nonprescription ibuprofen) over 6, 12, 24, and 48 hours after the first dose of study drug were calculated.
Time Frame: 6, 12, 24, and 48 hours
Population: The FAS included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TV-46763 5.0 mg/325 mg | TV-46763 7.5 mg/325 mg | TV-46763 10.0 mg/325 mg
Number analyzed (Participants) | 142 | 142 | 141 | 142
Participants
  Rescue medication use over 6 hours | 101 | 76 | 74 | 62
  Rescue medication use over 12 hours | 124 | 96 | 98 | 84
  Rescue medication use over 24 hours | 132 | 101 | 107 | 93
  Rescue medication use over 48 hours | 132 | 106 | 110 | 99

11. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious AEs. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: Day 1 up to Day 13
Population: The safety analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TV-46763 5.0 mg/325 mg | TV-46763 7.5 mg/325 mg | TV-46763 10.0 mg/325 mg
Number analyzed (Participants) | 142 | 142 | 141 | 142
Participants | 56 | 79 | 87 | 106

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 13
Description: The safety analysis set included all randomized participants who received at least 1 dose of study drug.
Arm/Group | Placebo | TV-46763 5.0 mg/325 mg | TV-46763 7.5 mg/325 mg | TV-46763 10.0 mg/325 mg
All-Cause Mortality (participants affected / at risk) | 0/142 | 0/142 | 0/141 | 0/142
Serious Adverse Events (participants affected / at risk) | 2/142 | 1/142 | 0/141 | 0/142
Other Adverse Events (participants affected / at risk) | 33/142 | 66/142 | 80/141 | 98/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=142) | TV-46763 5.0 mg/325 mg (N=142) | TV-46763 7.5 mg/325 mg (N=141) | TV-46763 10.0 mg/325 mg (N=142)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=142) | TV-46763 5.0 mg/325 mg (N=142) | TV-46763 7.5 mg/325 mg (N=141) | TV-46763 10.0 mg/325 mg (N=142)
Constipation (Gastrointestinal disorders) | 2 (2) | 26 (26) | 23 (23) | 30 (30)
Nausea (Gastrointestinal disorders) | 11 (12) | 37 (52) | 54 (63) | 68 (96)
Vomiting (Gastrointestinal disorders) | 4 (4) | 18 (24) | 27 (37) | 36 (67)
Alanine aminotransferase increased (Investigations) | 1 (1) | 9 (9) | 5 (5) | 5 (5)
Dizziness (Nervous system disorders) | 3 (4) | 10 (13) | 24 (26) | 23 (26)
Headache (Nervous system disorders) | 17 (22) | 13 (18) | 14 (16) | 24 (28)
Somnolence (Nervous system disorders) | 1 (1) | 8 (8) | 7 (7) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (3) | 5 (5) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.